CLINICAL TRIAL: NCT03436693
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate Efficacy and Safety of Canagliflozin (TA-7284) in Patients With Diabetic Nephropathy
Brief Title: Efficacy and Safety of Canagliflozin (TA-7284) in Patients With Diabetic Nephropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TA-7284-14
Record Dates: First submitted 2018-02-01; First posted 2018-02-19 (Actual); Results first posted 2024-07-15 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Diabetic Nephropathy
Keywords: Diabetic Nephropathy; Canagliflozin; Canaglu; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 2 | interventions — Canagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Canagliflozin 100mg (Experimental)
  Interventions: Drug: Canagliflozin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Canagliflozin — Canagliflozin 100mg orally once daily
  Other Names: TA-7284, Canaglu
  Arms: Canagliflozin 100mg
Drug: Placebo — Placebo orally once daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Canagliflozin (TA-7284) in Japanese patients with Diabetic Nephropathy, compared with placebo

ELIGIBILITY:
Inclusion Criteria:

Additional criteria check may apply for qualification:

* Glycated hemoglobin(HbA1c) of ≥6.5% and ≤12.0%
* eGFR of ≥30 mL/min/1.73m2 and <90 mL/min/1.73m2
* The median UACR of the first morning void urine samples is ≥300 mg/g Cr and ≤5000 mg/g Cr
* Patients who are taking on angiotensin-converting enzyme inhibitor (ACE-I) or angiotensin receptor blocker (ARB)
* Patients who are under dietary management and taking therapeutic exercise for diabetes

Exclusion Criteria:

Additional criteria check may apply for qualification:

* Type I diabetes, diabetes mellitus resulting from pancreatic disorder, or secondary diabetes
* A diagnosis of non-diabetic renal disease
* Hereditary glucose-galactose malabsorption or primary renal glucosuria
* Class IV heart failure symptoms according to New York Heart Association (NYHA) functional classification
* Severe hepatic disorder or severe renal disorder
* Blood potassium level >5.5 mmoL/L
* Stable blood pressure (diastolic blood pressure (DBP) ≥100mmHg or systolic blood pressure (SBP) ≥180mmHg)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Tanabe Pharma Corporation
Locations (26):
- Japan (26):
  - Research site, Aichi
  - Research site, Chiba
  - Research site, Fukuoka
  - Research site, Fukushima
  - Research site, Gunma
  - Research site, Hiroshima
  - Research site, Hokkaido
  - Research site, Hyōgo
  - Research site, Ibaraki
  - Research site, Kagawa
  - Research site, Kagoshima
  - Research site, Kanagawa
  - Research site, Kumamoto
  - Research site, Mie
  - Research site, Nagano
  - Research site, Nagasaki
  - Research site, Okinawa
  - Research site, Osaka
  - Research site, Ōita
  - Research site, Saitama
  - Research site, Shizuoka
  - Research site, Tochigi
  - Research site, Tokyo
  - Research site, Wakayama
  - Research site, Yamagata
  - Research site, Yamaguchi

REFERENCES:
- [Result] Wada T, Mori-Anai K, Takahashi A, Matsui T, Inagaki M, Iida M, Maruyama K, Tsuda H. Effect of canagliflozin on the decline of estimated glomerular filtration rate in chronic kidney disease patients with type 2 diabetes mellitus: A multicenter, randomized, double-blind, placebo-controlled, parallel-group, phase III study in Japan. J Diabetes Investig. 2022 Dec;13(12):1981-1989. doi: 10.1111/jdi.13888. Epub 2022 Aug 9. PMID 35861630
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818

RESULTS

PARTICIPANT FLOW:
Groups:
- Canagliflozin 100mg: Canagliflozin 100mg orally once daily for 104 Weeks
- Placebo: Placebo orally once daily for 104 Weeks
Period: Overall Study
Arm/Group | Canagliflozin 100mg | Placebo
Started | 154 | 154
Completed | 124 | 127
Not Completed | 30 | 27
Not completed — Adverse Event | 22 | 10
Not completed — Physician Decision | 3 | 3
Not completed — Withdrawal by Subject | 4 | 13
Not completed — Progressive Disease | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Canagliflozin 100mg | Placebo | Total
Number analyzed (Participants) | 154 | 154 | 308
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (10.5) | 62.4 (11.1) | 62.5 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 25 | 64
  Male | 115 | 129 | 244
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian(Japanese) | 154 | 154 | 308

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With 30% Decline in Estimated Glomerular Filtration Rate (eGFR) From Baseline at Week 104
Description: Percentage of participants with 30% decline in eGFR was calculated by multiple imputation method for missing data.
Time Frame: Week 104
Population: Full Analysis Set. All Patients were analyzed according to their randomized treatment assignment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Canagliflozin 100mg | Placebo
Number analyzed (Participants) | 154 | 154
Percentage of Participants | 18.2 [11.7 to 24.8] | 29.5 [21.9 to 37.2]
Statistical Analysis 1: Comparison: Canagliflozin 100mg vs Placebo; Test type: Other — Point Estimate; Difference(Multiple imputation method) = 11.3, 95% CI 2-sided [1.2 to 21.5]

2. Secondary Outcome: Percentage of Participants With 40% Decline in eGFR From Baseline at Week 104
Description: Percentage of participants with 40% decline in eGFR was calculated by multiple imputation method for missing data.
Time Frame: Week 104
Population: Full Analysis Set. All Patients were analyzed according to their randomized treatment assignment.
Measure: Number (95% Confidence Interval); unit: percentage of Participants
Arm/Group | Canagliflozin 100mg | Placebo
Number analyzed (Participants) | 154 | 154
percentage of Participants | 10.1 [5.0 to 15.3] | 13.9 [8.0 to 19.9]
Statistical Analysis 1: Comparison: Canagliflozin 100mg vs Placebo; Test type: Other — Point Estimate; Difference(Multiple imputation method) = 3.8, 95% CI 2-sided [-4.1 to 11.7]

3. Secondary Outcome: Change From Baseline in eGFR at Week 104
Time Frame: Baseline and Week 104
Population: For Canagliflozin 100mg, Outcome measure for 30 patients was not assessed at a certain timepoint due to dropout.
  For Placebo, Outcome measure for 27 patients was not assessed at a certain timepoint due to dropout.
Measure: Least Squares Mean (Standard Error); unit: mL/min/1.73m^2
Arm/Group | Canagliflozin 100mg | Placebo
Number analyzed (Participants) | 124 | 127
mL/min/1.73m^2 | -10.39 (0.83) | -11.49 (0.83)
Statistical Analysis 1: Comparison: Canagliflozin 100mg vs Placebo; Test type: Superiority; p = 0.351, Mixed Models Analysis; Difference of LSMean = 1.09, 95% CI 2-sided [-1.21 to 3.40]

4. Secondary Outcome: Composite Endpoint of End-stage Renal Disease (ESRD), Doubling of Serum Creatinine, Renal Death, and Cardiovascular (CV) Death
Time Frame: up to approximately 108 weeks
Population: Full Analysis Set. All Patients were analyzed according to their randomized treatment assignment.
Measure: Number; unit: Event rate per 1000 patient-years
Arm/Group | Canagliflozin 100mg | Placebo
Number analyzed (Participants) | 154 | 154
Event rate per 1000 patient-years | 24.29 | 38.66
Statistical Analysis 1: Comparison: Canagliflozin 100mg vs Placebo; Test type: Superiority; p = 0.293, Regression, Cox; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.23 to 1.55]

5. Secondary Outcome: Change From Baseline in Percentage of Urine Albumin-to -Creatinine Ratio (UACR) at Week 104
Time Frame: Baseline and Week 104
Population: Canagliflozin 100mg: Outcome measure for 30 patients was not assessed at a certain timepoint due to dropout.
  Placebo: Outcome measure for 27 patients was not assessed at a certain timepoint due to dropout.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Canagliflozin 100mg | Placebo
Number analyzed (Participants) | 124 | 127
percent change | 0.612 [0.525 to 0.714] | 1.178 [1.010 to 1.373]
Statistical Analysis 1: Comparison: Canagliflozin 100mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Ratio of Geometric LSMean = 0.52, 95% CI 2-sided [0.418 to 0.646]

ADVERSE EVENTS:
Time Frame: up to approximately 108 weeks
Arm/Group | Canagliflozin 100mg | Placebo
All-Cause Mortality (participants affected / at risk) | 4/154 | 2/154
Serious Adverse Events (participants affected / at risk) | 43/154 | 33/154
Other Adverse Events (participants affected / at risk) | 106/154 | 106/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canagliflozin 100mg (N=154) | Placebo (N=154)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 2
Myocardial infarction (Cardiac disorders) | 6 | 1
Prinzmetal angina (Cardiac disorders) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1
Cataract (Eye disorders) | 9 | 2
Cataract cortical (Eye disorders) | 1 | 0
Diabetic retinopathy (Eye disorders) | 3 | 0
Glaucoma (Eye disorders) | 3 | 0
Retinal haemorrhage (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1
Duodenal perforation (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 2
Large intestine polyp (Gastrointestinal disorders) | 2 | 1
Pancreatic fistula (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 1 | 1
Gait disturbance (General disorders) | 1 | 0
Cholangitis sclerosing (Hepatobiliary disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Enteritis infectious (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Failure to anastomose (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal cord injury (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain stem infarction (Nervous system disorders) | 0 | 1
Facial paralysis (Nervous system disorders) | 1 | 0
Myelopathy (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Thalamus haemorrhage (Nervous system disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Bladder mass (Renal and urinary disorders) | 0 | 1
Diabetic nephropathy (Renal and urinary disorders) | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 2
Renal failure (Renal and urinary disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Canagliflozin 100mg (N=154) | Placebo (N=154)
Diabetic retinopathy (Eye disorders) | 9 | 10
Constipation (Gastrointestinal disorders) | 15 | 10
Diarrhoea (Gastrointestinal disorders) | 7 | 10
Oedema peripheral (General disorders) | 1 | 9
Bronchitis (Infections and infestations) | 8 | 10
Influenza (Infections and infestations) | 9 | 10
Nasopharyngitis (Infections and infestations) | 54 | 57
Contusion (Injury, poisoning and procedural complications) | 10 | 9
Skin abrasion (Injury, poisoning and procedural complications) | 3 | 8
Blood glucose decreased (Investigations) | 27 | 23
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 9
Dyslipidaemia (Metabolism and nutrition disorders) | 8 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 33 | 32
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 5 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 17
Diabetic nephropathy (Renal and urinary disorders) | 5 | 8
Eczema (Skin and subcutaneous tissue disorders) | 8 | 6
Hypertension (Vascular disorders) | 9 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-04-17): https://cdn.clinicaltrials.gov/large-docs/93/NCT03436693/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/93/NCT03436693/SAP_001.pdf